CLINICAL TRIAL: NCT06352541
Title: Phase I Clinical Study, Evaluating Safety and Tolerability of PRO-232 an Ophthalmic Solution, Versus Placebo, When Applied to the Ocular Surface of Ophthalmologically and Clinically Healthy Volunteers.
Brief Title: Study Evaluating PRO-232 an Ophthalmic Solution Compared to Placebo.
Acronym: PRO-232
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOPH232-0824/I
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Phase I, controlled, comparative, parallel groups, double blind, one center.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-232 (Experimental): * PRO-232. Moxifloxacin 0.5% y Dexamethasone Phosphate 0.1% Ophthalmic solution.
  * Dosage: 1 drop QID [4] (four times per day) for 7 days on right eye.
  Interventions: Drug: PRO-232
- Placebo (Placebo Comparator): * Placebo. Sodium Chloride.
  * Dosage: 1 drop QID [4] (four times per day) for 7 days on right eye.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PRO-232 — Moxifloxacin 0.5% and Dexamethasone Phosphate 0.1%
  Arms: PRO-232
Other: Placebo — Vehicle Control, ophthalmic solution
  Arms: Placebo

SUMMARY:
This is a phase I study evaluating safety and tolerability through the incidence of unexpected adverse events and IOP measurement, as well as through the incidence of stinging after its administration, compared to placebo.

DETAILED DESCRIPTION:
The variables to be evaluated include:

Primary (safety):

* Unexpected adverse events
* IOP

Primary (tolerability):

- Stinging

Secondary (safety):

* Expected and related adverse events
* BCVA
* Ocular surface stining

Secondary (tolerability):

- Other ocular symptoms (foreign body sensation and tearing)

The operational definition states a difference under 15% in order to consider non inferior the safety and tolerability profile of PRO-232 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to voluntarily give their signed informed consent.
* Ophthalmologically and clinically healthy subjects.
* Being able to and willing to comply with scheduled visits, treatment plan, and other study procedures.
* Age between 18 to 45 years.
* Male or female gender.
* Women of childbearing potential who have not undergone Bilateral Tubal Occlusion (BTO [Tubal Ligation]), hysterectomy, or bilateral oophorectomy must ensure continuation (initiated ≥ 30 days prior to signing the informed consent form [ICF]) of the use of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* Best corrected visual acuity (BCVA) of 20/30 or better in both eyes.
* Corneal staining ≤ grade I on the Oxford Scale.
* Having an intraocular pressure ≥ 10 and ≤ 21 mmHg.

Exclusion Criteria:

* History of hypersensitivity to fluoroquinolones, steroid anti-inflammatories, or any of the components of the drugs under investigation.
* Use of ophthalmic medications from any pharmacological group.
* Use of medications by any other route of administration.
* Use of non-steroidal anti-inflammatory drugs, steroid anti-inflammatory drugs, or antibiotics by any route of administration in the last 30 days.
* History of eye surgery in the last 6 months.
* Use of contact lenses for a period less than two weeks prior to the start of the study, and during the intervention period of this study.
* In the case of women: being pregnant, breastfeeding, or planning to become pregnant within the study period.
* Having participated in any clinical research study 30 days prior to inclusion in this study.
* Having previously participated in this same study.
* History of any chronic-degenerative disease, including Diabetes Mellitus or Systemic Arterial Hypertension.
* Diagnosis of glaucoma or ocular hypertension.
* Known diagnosis of liver or heart disease.
* Presenting active inflammatory or infectious disease at the time of entry into the study.
* Presenting unresolved lesions or traumas at the time of entry into the study.
* Having been subjected to non-ophthalmological surgical procedures in the last 3 months.
* Being or having an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is an employee of the research site or the sponsor, and who directly participates in this study.
* Active smoking (specified as the consumption of cigarettes regardless of the amount and frequency, 4 weeks prior to study inclusion and during the intervention period of this study).
* Active alcoholism (specified as the consumption of alcoholic beverages, regardless of the amount and frequency, 72 hours prior to study inclusion and during the intervention period of this study).

Elimination Criteria

* Withdrawal of their consent to participate in the study (informed consent form).
* Occurrence of a serious adverse event, whether related or not to the interventions, that in the opinion of the principal investigator (PI) and/or the sponsor, could affect the patient's fitness to safely continue with the study procedures.
* Non-tolerability or hypersensitivity to any of the compounds used during the tests -(fluorescein, tetracaine).
* Non-tolerability or hypersensitivity to any of the drugs under investigation.
* Adherence < 80% determined by the subject's diary and corroborated by the final weight of the research products (RP) compared to the initial weight.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence Unexpected Related Adverse Reactions | Days 0 (Basal Visit) 3 (Visit 1), 8 (Final Visit) and 12 (Safety Call)
  Any unfavorable medical condition affecting the subject after the administration of the investigation product, related to such intervention.
Changes in intraocular pressure (IOP) | Days 0 (Basal Visit) 3 (Visit 1), 8 (Final Visit)
  Previous instillation of topical anesthetic, the IOP (right eye) will be measured through a Goldmann tonometer during visits
Incidence of Stinging | Days 0 (Basal Visit, 3 (Visit 1) and 8 (Final Visit)
  The subjects will be questioned regarding this symptom's incidence (right eye), frecuency, duration and severity will not be considered, only its incidence will.

SECONDARY OUTCOMES:
Incidence of Expected Related Adverse Events | Days 0 (Basal Visit), 3 (Visit 1), 8 (Final Visit) and 12 (Safety Call)
  Incidence of expexted related adverse events according to those previously described in bibliography: itching, blurry vision, eyelid pain, conjunctival hyperemia, ocular hypertension.
Changes in Best Corrected Visual Acuity (BCVA) | Days 0 (Basal Visit), Days 3 (Visit 1) and 8 (Final Visit)
  BCVA will be evaluated through Snellen chart
Changes in the integrity of the ocular surface (fluorescein staining) | Days 0 (Basal Visit), Days 3 (Visit 1) and 8 (Final Visit)
  Changes in the integrity of the ocular surface using fluorescein staining and evaluated through the Oxford scale. The standard Oxford scale for fluorescein staining has the following criteria: Grade 0- Equal to or less than panel A; Grade I- Equal to or less than panel B, greater than panel A; Grade II- Equal to or less than panel C, greater than panel B; Grade III- Equal or less than panel D, greater than panel C; Grade IV- Equal or less than panel E, greater than panel D; Grade V- Greater than panel E.
Incidence of ocular symptoms (foreign body sensation and tearing) | Days 0 (Basal Visit), 3 (Visit 1), 8 (Final Visit)
  The subjects will be questioned regarding this symptoms' incidence.

IPD SHARING:
Plan to Share IPD: No